CLINICAL TRIAL: NCT00931008
Title: A Randomized, Double-Blind, Two-Way Crossover, Bioequivalence Study of SID530 and Taxotere® in Study Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer After Platinum Therapy Failure or Study Participants With Locally Advanced or Metastatic Breast Cancer Who Have Failed At Least One Prior Chemotherapeutic Regimen
Brief Title: Study to Evaluate SID 530 Compared to Taxotere
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SID530_2009
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2010-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Locally Advanced or Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SID530; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- SID530 (Experimental): Study participants who meet eligibility criteria will be randomized to one of two treatment sequences, SID530 or Taxotere (i.e., SID530 on Day 1 followed by Taxotere on Day 21 or Taxotere on Day 1 followed by SID530 on Day 21)
  Interventions: Drug: SID530, Taxotere
- Taxotere (Active Comparator): Study participants who meet eligibility criteria will be randomized to one of two treatment sequences, SID530 or Taxotere (i.e., SID530 on Day 1 followed by Taxotere on Day 21 or Taxotere on Day 1 followed by SID530 on Day 21)
  Interventions: Drug: SID530, Taxotere

INTERVENTIONS:
Drug: SID530, Taxotere — 75mg/m2

SUMMARY:
This is a multi-center, randomized, blinded, two-period, two-sequence, crossover study, with a minimum 3-week washout period between treatments.The study is designed to evaluate the bioequivalence of SID530 to Taxotere.

It will be conducted in study participants with locally advanced or metastatic NSCLC who have failed platinum therapy and also in participants with locally advanced or metastatic breast cancer who have failed at least one line of chemotherapy.

Eligible study participants must be planning to have at least two consecutive 21-day cycles with 75 mg/m2 docetaxel monotherapy.

The duration of study participation will be approximately 7 weeks. The study has three study phases: Screening (<=1 week), Cycle 1 (21 days), and Cycle 2 (21 days).

DETAILED DESCRIPTION:
Study participants who meet eligibility criteria will be randomized to one of two treatment sequences (i.e., SID530 on Day 1 followed by Taxotere on Day 21 or Taxotere on Day 1 followed by SID530 on Day 21). Randomization will be stratified by whether the study participant received prior docetaxel treatment.

All study participants will be premedicated with oral dexamethasone, 16 mg per day (e.g. 8 mg b.i.d.) for three days, starting one day prior to each study drug infusion, in order to reduce the incidence and severity of fluid retention as well as the severity of hypersensitivity reactions. During each treatment cycle, both the test and the reference treatments will receive identical dosages of docetaxel (i.e., 75 mg/m2, by i.v. infusion, over 1 hour).

Study completion will be defined as completing all protocol-specified procedures. Study participants who are prematurely withdrawn from the study will be requested to complete the assessments conducted at the Final Visit.

Blood samples for pharmacokinetic analysis will be obtained at the predefined times during Cycle 1 and Cycle 2.

Adverse events will be assessed throughout the study, including 21 days after the last study drug infusion. Hematology assessments,other laboratory parameters and vital signs will be assessed.

ELIGIBILITY:
Inclusion Criteria:Study participants

* Has provided written informed consent
* Is at least 18 years of age
* Has histologically or cytologically confirmed non-small cell lung (NSCLC) or breast cancer (BC) that is locally advanced or metastatic
* Has at least two planned consecutive 21-day cycles with 75 mg/m2 docetaxel monotherapy
* Has a life expectancy of at least 3 months
* Has Eastern Cooperative Oncology Group Performance Scale (ECOG PS) is in the range of 0-2 at the time of randomization
* Has the Proper laboratory values within 1 week prior to randomization
* Has negative serum pregnancy test within 1 week before first study drug administration (for women of childbearing potential, only)
* Is willing to practice medically accepted contraception (if the risk of conception exists) throughout the study period (from Screening until the Final Visit)

Exclusion Criteria:Study participants

* Has had any chemotherapy within 4 weeks before date of first study treatment
* Has experienced severe side effects from (or severe hypersensitivity to) prior docetaxel treatment (or other drugs formulated with polysorbate 80, hydroxypropylbetadex, or povidone) such that discontinuation of the treatment was required
* Has a history of hypersensitivity to dexamethasone
* Is pregnant, lactating, or breastfeeding
* Is taking one or more compounds that induce, inhibit, or are metabolized by cytochrome P450 3A4
* Has had treatment in another clinical study within the past 30 days
* Has medical or psychological conditions that would not permit the study participant to complete the study or sign informed consent
* Is unlikely to comply with the protocol requirements, instructions and study-related restrictions
* Has any other disease, dysfunction (including alcohol or drug abuse), physical examination or laboratory finding which, in the investigator's opinion, would exclude the participant from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
to test the bioequivalence of SID530 (test) to Taxotere | 7 weeks

SECONDARY OUTCOMES:
to evaluate the of safety and tolerability of SID530 as compared to the marketed Taxotere. | 7 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Advanced Clinical Research Pharma, Miami, Florida
  - Gabrail Cancer Center, Canton, Ohio
- India (2):
  - City Cancer Hospital, Vijayawada AndhraPradesh, Ch. Venkatka Krishnayya
  - Kamakshi Memorial Hospital, No-1, Radial Road, Pallikarani, Chennai, Tamilnadu